CLINICAL TRIAL: NCT03952364
Title: The PRECIOUS Study: Predicting Crohn's & ColitIs Outcomes in the United States
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: PredictImmune Ltd (Industry)
Collaborators: Crohn's and Colitis Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: The Precious Study
Record Dates: First submitted 2019-05-14; First posted 2019-05-16 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Crohn Disease; Ulcerative Colitis; IBD; Inflammatory Bowel Diseases
Keywords: Crohn's Disease; Ulcerative Colitis; IBD; Inflammatory Bowel Disease; Precious
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Following patient consent and recruitment to the study, a 2.5 ml blood sample will be collected in a PAXgene tube.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: PredictSURE IBD™ — To evaluate a test called PredictSURE IBD™ in the US population

SUMMARY:
A multi-center observational study based at referral centers and community hospitals within the US. Patients' blood will be collected at enrollment for testing with PredictSURE IBD™, which will occur at a later date. Patients will be prospectively followed up for 12 months with clinicians treating according to local standard of care, with a step-up or accelerated step-up regimen. Clinicians and patients will be blinded to the biomarker results.

DETAILED DESCRIPTION:
This is a multi-center, observational study of newly diagnosed IBD (CD or UC) patients. The Study aims to assess whether a prognostic biomarker can stratify IBD patients in the US.

ELIGIBILITY:
Inclusion Criteria:

* Active UC or CD with typical symptoms in conjunction with at least one objective measure of disease activity: elevated CRP, calprotectin, endoscopic evidence.
* Not currently receiving systemic therapy* with steroids, immunomodulators or biologics, and at least 7 days since the last steroid dose.
* Due to be managed using a "step-up" or "accelerated step-up" approach (so will not receive biologics as first line therapy).
* Aged 16-80 years old.

Note, the ideal patients for this study are newly diagnosed patients who are treatment-naïve.

Exclusion Criteria:

* The presence of any of the following will preclude patient inclusion:
* Patients with fistulating peri-anal Crohn's disease or active perianal sepsis.
* Obstructive symptoms and evidence of a fixed stricture on radiology or colonoscopy.
* Patients who are scheduled to start on "top-down" therapy or receive biologics as a first line therapy

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The target patient populations are newly diagnosed, active CD or UC in patients who are immunomodulator and anti-TNFα treatment naïve.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-10-10 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
To stratify patients at diagnosis into high and low- risk cohorts | 12 month follow up
  Stratifying patients into high or low risk of following an aggressive disease course requiring frequent treatment escalations.

CONTACTS AND LOCATIONS:
Overall Officials: James Lee, MD, Principal Investigator — PredictImmune Ltd
Locations (8):
- United States (8):
  - University of Miami Crohn's and Colitis Center, Miami, Florida
  - Washington University in St. Louis, St Louis, Missouri
  - Rutgers Robert Wood Johnson Medical School (Adult), New Brunswick, New Jersey
  - Rutgers Robert Wood Johnson Medical School (Prediatric), New Brunswick, New Jersey
  - Manhattan Clinical Research, LLC., New York, New York
  - NYU Langone Health, New York, New York
  - Weill Cornell Medical Center, New York, New York
  - ClinSearch, Chattanooga, Tennessee

IPD SHARING:
Plan to Share IPD: No